CLINICAL TRIAL: NCT04261036
Title: Vitamin C for the Prevention of Catheter-associated Urinary Tract Infections in Women Who Undergo Elective Gynecological Surgeries: a Study Protocol for a Randomized Double Blinded Controlled Trial.
Brief Title: Vitamin C for the Prevention of UTI in Women Who Undergo Elective Gynecological Surgeries
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unfortunately, the economic crisis in Lebanon precluded utilization of available funding to recruit patients at the specified institution. No patients were recruited.
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Tony Bazi, Associate Professor of Clinical Obstetrics and Gynecology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OGY.TB.09/BIO-2017-0609
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Catheter-Associated Urinary Tract Infection, Ascorbic Acid
Keywords: Vitamin C; CAUTI; Ascorbic Acid
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Vitamin C and Placebo pills will be blindly labeled and assorted in opaque containers in the Pharmacy department according to a computer generated list that allocated random assignment of vitamin C or placebo to a 200 positions (serial numbers from 1 to 200).
  The research assistant in charge of the recuitment will not be aware of the content of each opaque container and would be providing them to patients according to the order in which they are recruited starting with container number 1, then 2 and so on.
  The primary care provider and the investigators are blinded as well as they are not aware of the assignment of each recruited patient to placebo vs interventional arm.
  It is only upon completion of data collection that results would be compared with the randomized generated list in order to link the recruited patients and their collected data with their original assignment to placebo vs intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Women on a vitamin C regimen (Experimental): Women who are undergoing elective gynecological surgeries and who are randomized to take 1g of vitamin C for 14 days.
  Interventions: Drug: Ascorbic Acid 1000 mg
- Women on a placebo regimen (Placebo Comparator): Women who are undergoing elective gynecological surgeries and who are randomized to take placebo for 14 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ascorbic Acid 1000 mg — 1000 mg ascorbic acid (Vitamin C) for 14 days post-op after an elective gynecological surgery.
  Arms: Women on a vitamin C regimen
Other: Placebo — Placebo pills for 14 days post-op after an elective gynecological surgery.
  Arms: Women on a placebo regimen

SUMMARY:
This open-label randomized trial aims at assessing the role of Vitamin C pills in the prevention of catheter-associated urinary tract infections in women undergoing elective gynecological surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant women at least 18 years of age visiting the Preadmission unit (PAU) or the OBGYN floor (7N), presenting for elective GYN surgery at the American University of Beirut Medical Center (AUBMC).

Exclusion Criteria:

* Any women with the following:

  1. Nephrolithiasis
  2. Congenital anomaly or neurogenic bladder
  3. Allergy to ascorbic acid
  4. Who require therapeutic anticoagulant medicine during the 6 weeks after surgery
  5. Surgery did involve a fistula repair or a vaginal mesh removal
  6. Positive Urinalysis in the PAU
  7. Recurrent UTI's
  8. Diabetes
  9. G6PD
  10. Hemochromatosis
  11. Renal disorders

Patients already taking Vitamin C supplementation will also be excluded from the study.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who experienced clinically diagnosed and treated UTI. | 14 days
  Urinary tract infection is diagnosed by a positive urine culture.

SECONDARY OUTCOMES:
Proportion of participants with asymptomatic bacteruria | 14 days
  Participants with positive urine culture but no symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foxman B, Cronenwett AE, Spino C, Berger MB, Morgan DM. Cranberry juice capsules and urinary tract infection after surgery: results of a randomized trial. Am J Obstet Gynecol. 2015 Aug;213(2):194.e1-8. doi: 10.1016/j.ajog.2015.04.003. Epub 2015 Apr 13. PMID 25882919
- [Background] Ochoa-Brust GJ, Fernandez AR, Villanueva-Ruiz GJ, Velasco R, Trujillo-Hernandez B, Vasquez C. Daily intake of 100 mg ascorbic acid as urinary tract infection prophylactic agent during pregnancy. Acta Obstet Gynecol Scand. 2007;86(7):783-7. doi: 10.1080/00016340701273189. PMID 17611821
- [Background] Carlsson S, Wiklund NP, Engstrand L, Weitzberg E, Lundberg JO. Effects of pH, nitrite, and ascorbic acid on nonenzymatic nitric oxide generation and bacterial growth in urine. Nitric Oxide. 2001 Dec;5(6):580-6. doi: 10.1006/niox.2001.0371. PMID 11730365
- [Background] Trautner BW, Darouiche RO. Catheter-associated infections: pathogenesis affects prevention. Arch Intern Med. 2004 Apr 26;164(8):842-50. doi: 10.1001/archinte.164.8.842. PMID 15111369
- [Background] Barbosa-Cesnik C, Brown MB, Buxton M, Zhang L, DeBusscher J, Foxman B. Cranberry juice fails to prevent recurrent urinary tract infection: results from a randomized placebo-controlled trial. Clin Infect Dis. 2011 Jan 1;52(1):23-30. doi: 10.1093/cid/ciq073. PMID 21148516
- [Background] Hickling DR, Nitti VW. Management of recurrent urinary tract infections in healthy adult women. Rev Urol. 2013;15(2):41-8. PMID 24082842
- [Background] Wald HL, Ma A, Bratzler DW, Kramer AM. Indwelling urinary catheter use in the postoperative period: analysis of the national surgical infection prevention project data. Arch Surg. 2008 Jun;143(6):551-7. doi: 10.1001/archsurg.143.6.551. PMID 18559747